CLINICAL TRIAL: NCT04697030
Title: Behavioral Outcomes Among Adolescent Population During Covid-19 Pandemic Lockdown in Pakistan: A Lower Middle Income Country Experience
Brief Title: Burnout Among Adolescent Population During Covid-19 Lockdown in Pakistan
Status: Completed | Type: Observational
Sponsor: Sialkott College of Physical Therapy (Other)
Responsible Party: Principal Investigator, Wajida Perveen, Head of Physical Therapy Department., Sialkott College of Physical Therapy
Other Study IDs: 129-2020
Record Dates: First submitted 2020-12-31; First posted 2021-01-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Burnout, Psychological; Covid-19 Pandemic
Keywords: adolescent Population; Covid-19 Pandemic; Burnout; Mental Health
MeSH Terms: conditions — Burnout, Psychological; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The lethal severe acute respiratory syndrome coronavirus 2 (SARS-COV2) which caused the COVID-19 pandemic starting at the end of 2019 has affected the lives of children and adolescents globally. world adopted the lockdown to prevent spread of the infection and protect the population. lockdown suspended out of home activities of almost everyone, along with health benefits, yielding some side effects as well including burnout. The burnout includes physical and emotional burnout, physical burnout refers to the lack of interest in any physical activity to the point of a rebel and the emotional burnout of teenagers refers to a syndrome including features such as behavior changes, thinking change, feeling change, health change leading to stress and other pathological disturbances. Together the external and internal factors lead to overall personality destruction.

It was an observational study with a sample size of 443 participants.

DETAILED DESCRIPTION:
Objective of the study was to analyze the change in behavioral patterns, its impact, and peer pressure caused by lockdown during Pandemic COVID-19 among the adolescent population of Sialkot Pakistan.

It was an observational study with a sample size of 443 participants. The study was conducted after ethical approval by Institutional Review Board, Sialkot college of Physical Therapy wide Reference no. SCPT-IRB-DPT-129-2020 dated 01-09-2020. Data were collected from different institutions in Sialkot, Pakistan. The target population of our study was adolescents of age 13-19 years. Regression analysis was done to find the predictor factors mobile use and COVID-19 lockdown on the dependent variable the Burnout score. The correlation was applied among mobile phone use, lockdown, and burnout score.

ELIGIBILITY:
Inclusion Criteria:

* students of the above age group who started to go to the school/ colleges/ university/Academies.
* those who consent to participate in the study.

Exclusion Criteria:

* students who were unable to visit their institution and stayed at home.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: this study was conducted on adolescent population of students.
Sampling Method: Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Burnout Rating Scale | data were collected within one month after six month stay at home during Covid-19 l-Lockdown.
  Burnout Rating Scale total score ranges from 0-50, the higher the score more will be the risk and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Wajida Perveen, MS-OMPT, Study Director — Sialkot College of Physical Therapy; Ijaz Amin, MS-Ortho, Study Chair — Sialkot College of Physical Therapy; Roha Asif, PhD*, Study Director — Sialkot College of Physical Therapy
Locations (1):
- Sialkot College of Physical Therapy, Amin Welfare & Teaching Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No